CLINICAL TRIAL: NCT02577731
Title: Hematopoietic Stem Cell Dysfunction in the Elderly After Severe Injury: Chronic Stress and Anemia Recovery Following Major Trauma
Brief Title: Hematopoietic Stem Cell Dysfunction in the Elderly After Severe Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB201601386-N; 1R01GM113945-01 (NIH); IRB 106-2013 (Other: Univeristy of Florida); 5R01GM105893 (NIH); OCR30562 (Other: University of Florida)
Record Dates: First submitted 2015-10-01; First posted 2015-10-16 (Estimated); Last update posted 2026-01-15 (Actual); Status verified 2025-04

CONDITIONS: Trauma Injury
Keywords: Trauma
MeSH Terms: conditions — Accidental Injuries; Wounds and Injuries | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Severe Trauma (Other): Bone marrow collection. Blood collection. Clinical data collection.
  Interventions: Other: Bone marrow collection; Other: Blood collection; Other: Clinical data collection
- Elective Hip Repair (Other): Bone marrow collection. Blood collection. Clinical data collection.
  Interventions: Other: Bone marrow collection; Other: Blood collection; Other: Clinical data collection
- Healthy Young Bone Marrow Control (Other): Deidentified freshly isolated bone marrow samples from healthy young control subjects will be purchased for a tissue bank.
  Interventions: Other: Bone marrow collection

INTERVENTIONS:
Other: Bone marrow collection — Bone marrow will be collected from the patient at time of orthopedic repair in the operating room. A second sample may be collected if the patient is required to return to the operating room for further repair of orthopedic injury.
Other: Blood collection — Blood sample collection will be collected from the patient at time of orthopedic repair in the operating room. A second sample may be collected if the patient is required to return to the operating room for further repair of orthopedic injury.
  Arms: Elective Hip Repair; Severe Trauma
Other: Clinical data collection — Clinical data collection will encompass demographic information, past and present medical records, laboratory, microbiology, and all other test results, x-ray, CT, MRI, US and all other imaging test results, records about any medication received during admission, records of physical exam during admission, records of all vital signs and hemodynamic monitoring during admission, records of any procedure or intervention during admission, records of any procedure or intervention during hospital admission, condition at the discharge and discharge facility.
  Arms: Elective Hip Repair; Severe Trauma

SUMMARY:
Traumatic injury is a leading cause of morbidity and mortality in young adults, and remains a substantial economic and health care burden. Despite decades of promising preclinical and clinical investigations in trauma, investigators understanding of these entities is still incomplete, and few therapies have shown success. During severe trauma, bone marrow granulocyte stores are rapidly released into the peripheral circulation. This release subsequently induces the expansion and repopulation of empty or evacuated space by hematopoietic stem cells (HSCs). Although the patient experiences an early loss of bone marrow myeloid-derived cells, stem cell expansion is largely skewed towards the repopulation of the myeloid lineage/compartment. The hypothesis is that this 'emergency myelopoiesis' is critical for the survival of the severely traumatized and further, failure of the emergency myelopoietic response is associated with global immunosuppression and susceptibility to secondary infection. Also, identifying the release of myeloid derived suppressor cells (MDSCs) in the circulation of human severe trauma subjects. This process is driven by HSCs in the bone marrow of trauma subjects. Additionally, MDSCs may have a profound effect on the nutritional status of the host. The appearance of these MDSCs after trauma is associated with a loss of muscle tissue in these subjects. This muscle loss and possible increased catabolism have huge effects on long term outcomes for these subjects. It is the investigator's goal to understand the differences that occur in these in HSCs and muscle cells as opposed to non-injured and non-infected controls. This work will lead to a better understanding of the myelopoietic and catabolic response following trauma.

DETAILED DESCRIPTION:
This is a prospective study to understand how trauma injuries changes the hematopoeitic stem cells (HSCs) in the bone marrow and muscle cells after trauma injury in elderly subjects is different when compared to non-injured subjects.

There will be three groups for this study: 1) Elective hip surgery subjects, 2) Trauma subjects and 3) deidentified bone marrow of healthy controls.

Samples of bone marrow and a blood sample will be collected at the time of surgery. The deidentified bone marrow of healthy controls will come from a tissue bank.

The blood will be used to perform PB colony assays, ELISAs to test for the following parameters: EPO, G-CSF, Reticulocyte, iron levels and cytokines and inflammatory markers.

The bone marrow and blood samples will be processed and sorted to isolate hematopoeitic stem cells for genomic content to determine genomic expression, oxidative stress, mitochondrial activity, apoptosis, autophagy, analysis of circulating erythroid progenitor cells, reticulocytes, granulocyte-colony stimulating factor assays, erythropoietin and iron levels.

Clinical data and hemodynamic measurements will be collected daily while subjects are hospitalized and trauma surgery subjects will be followed to evaluate for malunion and subsequent additional surgical procedures for repair.

ELIGIBILITY:
Severe Trauma Population

Inclusion criteria will be:

1. All adults (age ≥18 to 54)
2. Blunt and/or penetrating trauma resulting in long bone or pelvic fractures requiring ORIF or closed reduction percutaneous pinning (CRPP).
3. Blunt and/or penetrating trauma patient with either:

   1. hemorrhagic shock defined by: i. systolic BP (SBP) ≤ 90 mmHg or ii. mean arterial pressure≤ 65 mmHg or iii. base deficit (BD) ≥ 5 meq or iv. lactate ≥ 2
   2. Or injury severity score (ISS) greater than or equal to 15.
4. All adults (age 55 and older) require:

   1. Blunt and/or penetrating trauma resulting in log bone or pelvic fractures requiring ORIF or CRPP
   2. Either hemorrhagic shock defined by: i. Systolic BP (SBP) ≤ 90 mmHg or ii. Mean arterial pressure ≤ 65 mmHg or iii. Base deficit (BD) ≥5 meq or iv. Lactate ≥ 2
   3. Or Injury Severity Score (ISS) greater than or equal to 15.
5. Ability to obtain Informed Consent prior to OR repair of injury.

Exclusion Criteria will be:

1. Patients not expected to survive greater than 48 hours.
2. Prisoners.
3. Pregnancy.
4. Patients receiving chronic corticosteroids or immunosuppression therapies.
5. Previous bone marrow transplantation.
6. Patients with End Stage Renal Disease.
7. Patients with any pre-existing hematological disease.

Elective Hip Repair Population

Inclusion criteria will be:

1. All adults (age ≥18)
2. Patient undergoing elective hip repair for non-infectious reasons.
3. Ability to obtain Informed Consent prior to operation.

Exclusion Criteria will be:

1. Pregnancy.
2. Prisoners.
3. Patients receiving chronic corticosteroids or immunosuppression therapies.
4. History of receiving Chemotherapy or Radiation within the last 6 months
5. Previous bone marrow transplantation

7. Patients with End Stage Renal Disease 8. Patients with any pre-existing hematological disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2014-01 (Actual); Primary Completion 2026-12-28 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Analyze the genomics response of hematopoietic cells between the groups | Baseline
  Through negative isolation columns and flow sorting to isolate the hematopoietic stem cells (HSCs) from a sample for appropriate analysis. The sample will then be enriched using a lineage depletion column which will remove all mature hematopoietic cells. The HSCs will be phenotyped and sorted as CD34+ CD38- Thy1+ CD45RA-. HSCs will be lysed and the RNA genomic content will be isolated. The genomic content will then be processed onto a GeneChip® microarray to analyze the genomic expression.
Analyze the muscle dysfunction between the groups for oxidative stress | Baseline
Analyze the muscle dysfunction between the groups for mitochondrial activity | Baseline
Analyze the muscle dysfunction between the groups for apoptosis | Baseline
Analyze the muscle dysfunction between the groups for autophagy | Baseline

SECONDARY OUTCOMES:
The pathophysiology of injury-associated persistent anemia through PB colony assays of blood. | Baseline
The pathophysiology of injury-associated persistent anemia through ELISA test of blood. | Baseline

OTHER OUTCOMES:
Analyze the genomics response of hematopoietic cells between the groups at additional follow-up surgery | Approximately 8 months
  Through negative isolation columns and flow sorting to isolate the hematopoietic stem cells (HSCs) from a sample for appropriate analysis. The sample will then be enriched using a lineage depletion column which will remove all mature hematopoietic cells. The HSCs will be phenotyped and sorted as CD34+ CD38- Thy1+ CD45RA-. HSCs will be lysed and the RNA genomic content will be isolated. The genomic content will then be processed onto a GeneChip® microarray to analyze the genomic expression.
Analyze the muscle dysfunction between the groups at additional follow-up surgery for oxidative stress | Approximately 8 months
Analyze the muscle dysfunction between the groups at additional follow-up surgery for mitochondrial activity | Approximately 8 months
Analyze the muscle dysfunction between the groups at additional follow-up surgery for apoptosis | Approximately 8 months
Analyze the muscle dysfunction between the groups at additional follow-up surgery for autophagy | Approximately 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Philip Efron, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health Shands Hospital at the University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Derived] Munley JA, Willis ML, Gillies GS, Kannan KB, Polcz VE, Balch JA, Barrios EL, Wallet SM, Bible LE, Efron PA, Maile R, Mohr AM. Exosomal microRNA following severe trauma: Role in bone marrow dysfunction. J Trauma Acute Care Surg. 2024 Apr 1;96(4):548-556. doi: 10.1097/TA.0000000000004225. Epub 2023 Dec 28. PMID 38151766
- [Derived] Munley JA, Kelly LS, Gillies GS, Kannan KB, Pons EE, Bible LE, Efron PA, Mohr AM. EFFECTS OF TRAUMA PLASMA-DERIVED EXOSOMES ON HEMATOPOIETIC PROGENITOR CELLS. Shock. 2023 Apr 1;59(4):591-598. doi: 10.1097/SHK.0000000000002094. Epub 2023 Feb 16. PMID 36772985